CLINICAL TRIAL: NCT00883922
Title: Central Venous Saturation (ScvO2) Monitoring in Pediatric Patients Undergoing Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Aman Mahajan, Principal Investigator, University of California, Los Angeles
Other Study IDs: 06-12-078-03
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Congenital Heart Defects; Cardiac Surgery
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Children (ages 0-12) that have heart surgery are often at a high risk of developing complications and have to be continuously monitored. Part of the routine care at UCLA includes using a monitor (continuous central venous oxygen saturation-ScvO2) to measure the amount of oxygen saturation in the tissues (indirectly) during surgery and in the intensive care unit. However, there is not much data on the use and effectiveness of this monitor in comparison to other monitors used for children.

The purpose of this study is to further evaluate the effectiveness of the continuous central venous oxygen saturation (ScvO2) monitor in children and compare it with other monitors during a heart surgery. This is an observational study and the patients will not undergo any research specific procedures in the operating room (OR). The investigators will observe and record de-identified information, such as vital signs (heart rate, blood pressure, etc.), to evaluate the importance of the monitor. This study will also look at the demographics (age, gender, diagnosis, etc.) and treatments (type of surgery) received children undergoing heart surgery to improve quality of care. The investigators will also observe the same parameters in the ICU. The investigators hypothesized that low central venous saturations are associated with worse clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (age 0-12 years) scheduled for cardiac surgery and requiring placement of a central venous catheter.

Exclusion Criteria:

* Patients with contraindications for placement of a central venous catheter will be excluded from this study.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients scheduled for cardiac surgery
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States